CLINICAL TRIAL: NCT02692261
Title: Evaluation of Hyaluronic Matrix, Used With Xenograft, Efficacy in Sinus Augmentation by Histomorphometry and Micro Computed Tomography
Brief Title: Hyaluronic Matrix Efficacy for Maxillary Sinus Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, EZGİ DOĞAN, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-14030
Record Dates: First submitted 2016-02-17; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Sinus; Dental
MeSH Terms: conditions — Fistula | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyalossᵀᴹ matrix (Active Comparator): Each 0.5 cc Collagenated Heterolog Bone Graft, mixed with two bundles of Hyalossᵀᴹ matrix and a few drops of sterile saline solution used for maxillary sinus augmentation
  Interventions: Procedure: Maxillary Sinus Augmentation
- Apatos alone xenograft (Active Comparator): Each sinus was filled with 1 gr xenograft (with or without Hyaluronic Acide) for maxillary sinus augmentation
  Interventions: Procedure: Maxillary Sinus Augmentation

INTERVENTIONS:
Procedure: Maxillary Sinus Augmentation — Each 0.5 cc Collagenated Heterolog Bone Graft, mixed with two bundles of Hyalossᵀᴹ matrix and a few drops of sterile saline solution
  Other Names: Hyaloss matrix
Procedure: Maxillary Sinus Augmentation — Control group sinuses filled with heterolog bone graft alone

SUMMARY:
Sinus augmentation is a predictable method when alveolar bone height is not sufficient for dental implant placement in posterior maxillary alveolar region..The aim of this prospective, randomized, controlled clinical study is comparison of hyaluronic acid originated matrix and equine derived xenograft with only xenograft use in sinus augmentation by micro computed tomography and histomorphometry.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients
* Requiring bilateral maxillary sinus augmentation (residual crest height ≤ 4 mm)

Exclusion Criteria:

* Advanced systemic diseases
* Chronic medication use
* Maxillary sinus disease
* Current pregnancy
* Lactation
* Smoking habit

Ages: 33 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of newly formed bone calculated from bone biopsises by Micro-CT and Histomorphometry | 4 months after surgery
  Biological parameter obtained by analyzing bone biopsises

CONTACTS AND LOCATIONS:
Overall Officials: Feriha Caglayan, Professor, Study Chair — Hacettepe University

IPD SHARING:
Plan to Share IPD: No